CLINICAL TRIAL: NCT02887625
Title: Efficacy and Durability of Glucagon Like Peptide 1 Receptor Agonists (GLP-1 RA)/Thiazolidinedione Versus Basal Bolus Insulin Therapy in Poorly Controlled Type 2 Diabetic Patients (T2DM) Patients on Sulfonylurea Plus Metformin
Brief Title: Exenatide Plus Pioglitazone Versus Insulin in Poorly Controlled T2DM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr. Muhammad Abdulghani (Industry)
Responsible Party: Sponsor-Investigator, Dr. Muhammad Abdulghani, Professor of Medicine, Hamad Medical Corporation
Organization: Hamad Medical Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NPRP 5-273-3-079
Record Dates: First submitted 2016-08-16; First posted 2016-09-02 (Estimated); Last update posted 2016-09-02 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Exenatide; Insulin Glargine; Insulin Aspart

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Therapy (Experimental): pioglitazone (actos) 30 mg per day and exenatide (bydureon) 2 mg per week
  Interventions: Drug: Pioglitazone plus exenatide
- Insulin Therapy (Active Comparator): insulin glargine (lantus) will be started every morning and the dose will be weekly increase to achieve fasting plasma glucose (FPG) <110 mg/dl.
  and Aspart insulin will be started before meals and the dose is adjusted to maintain HbA1c <7.0% and postprandial plasma glucose (PPG) <140 mg/dl
  Interventions: Drug: insulin glargine and insulin aspart

INTERVENTIONS:
Drug: Pioglitazone plus exenatide — pioglitazone will be started at 30 mg/day and bydureon at 2 mg/week
  Other Names: actos and bydureon
  Arms: Combination Therapy
Drug: insulin glargine and insulin aspart — the dose will be escalated to maintain HbA1c <7.0%
  Other Names: lantus
  Arms: Insulin Therapy

SUMMARY:
To compare efficacy, safety and durability of combination therapy with pioglitazone plus GLP-1 RA versus basal bolus insulin in poorly controlled T2DM patients on metformin plus sulfonylurea

DETAILED DESCRIPTION:
poorly controlled (HbA1c >7.5%) T2DM patients (18-75 years of age) on maximal/near maximal dose of sulfonylurea plus metformin who otherwise are healthy will be randomized to receive:

1. exenatide weekly injection (2 mg/week)
2. glargine insulin plus insulin aspart which will be titrated to maintain HbA1c <7.0%

ELIGIBILITY:
Inclusion Criteria:

* T2DM poorly controlled (HbA1c >7.5%) on metformin (>1700 mg/day) plus sulfonylurea

Exclusion Criteria:

* type 1 diabetes (T1DM) patients receiving therapy with pioglitazone, GLP-1 RA and insulin abnormal kidney, liver or heart function patients with malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-05 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
HbA1c | 3 years
  difference in HbA1c between the two treatment groups will be compared at 1 and at 3 years to determine efficacy and durability of each treatment

SECONDARY OUTCOMES:
percentage of patients who achieve HbA1c <7.0% and <6.5% at 1 year and at 3 years | 3 years
hypoglycemia rate | 3 years
  will be measured as absolute event rate per patient year of follow up
change in the FPG | 3 years
  change in FPG from time zero to 1 year and from baseline to 3 years in each treatment group
change in body weight | 3 years
  change in body weight from time zero to 1 year and to 3 years in each treatment group

CONTACTS AND LOCATIONS:
Overall Officials: Amin Jayyousi, MD, Principal Investigator — HMC
Locations (1):
- Hamad General Hospital, Doha, Qatar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdul-Ghani M, Migahid O, Megahed A, Adams J, Triplitt C, DeFronzo RA, Zirie M, Jayyousi A. Combination Therapy With Exenatide Plus Pioglitazone Versus Basal/Bolus Insulin in Patients With Poorly Controlled Type 2 Diabetes on Sulfonylurea Plus Metformin: The Qatar Study. Diabetes Care. 2017 Mar;40(3):325-331. doi: 10.2337/dc16-1738. Epub 2017 Jan 17. PMID 28096223